CLINICAL TRIAL: NCT03908151
Title: Five and Ten Year Results of the CMK21 Hip System
Acronym: CMK21
Status: Terminated | Type: Observational
Why Stopped: Business Decision
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R11008-2B
Record Dates: First submitted 2016-08-26; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis
Keywords: hip prosthesis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CMK21 Hip system — Total hip arthroplasty

SUMMARY:
Five and ten year results of the CMK21 Hip system

DETAILED DESCRIPTION:
This study is being conducted to collect long term retrospective and prospective clinical and radiological data to evaluate the safety of revision rate and adverse events, and efficacy of clinical and patient assessment of the CMK21 hip stem in primary total hip arthroplasty.

ELIGIBILITY:
Inclusion:

* The patients enrolled in the study were already operated at the time of the screening.
* All the patients with osteoarthritis of the hip who received CMK21 hip stem between 2005 and 2007.
* Skeletally mature patients requiring primary total hip arthroplasty due to non-inflammatory arthritis (degenerative joint disease) such as osteoarthritis, avascular necrosis, or traumatic arthritis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all patients who received a CMK21 hip stem as part of a primary total hip arthroplasty between 2005 and 2007. This includes all diagnoses, all ages, male and female.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-12; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Implant revision rate | 5 years
  Listing of implant status at 5 years to analyse the survival rate
Implant revision rate | 10 years
  Listing of implants status at 10 years to analyse the survival rate
Device related adverse events | 10 years
  Medical chart will be reviewed and device related events collected to monitor the safety
Device related adverse events | 5 and 10 years
  Device related adverse events will be collected to monitor the safety
Radiographic assessment | 5 and 10 Years
  Radiolucent lines and radiosclerotic lines at both the bone cement and cement prosthesis interface
Radiographic assessment | 5 and 10 Years
  Position and fixation of the components
Radiographic assessment | 5 and 10 Years
  the occurrence of osteolysis
Radiographic assessment | 5 and 10 Years
  the occurrence of heterotopic bone formation
Radiographic assessment | 5 and 10 Years
  the occurrence of atrophy or hypertrophy
Radiographic assessment | 5 and 10 Years
  the occurrence of cement tears/fractures

SECONDARY OUTCOMES:
Harris Hip Score (HHS) | 5 and 10 years
  Harris Hip Score is a clinical evaluation which consists of a maximum of 100 points (best possible outcome) covering pain (1 item, 44 points), function (7 items 47 points total), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points total).
EuroQoL Five Dimensions Questionnaire (EQ-5D) | 5 and 10 years
  The EuroQoL Five Dimensions Questionnaire is a subject self-assessment of quality of life and consists of five questions covering the dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which subjects can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

CONTACTS AND LOCATIONS:
Overall Officials: Beate Hanson, VP, PhD, Study Chair — Vice President, Global Clinical Strategy
Locations (2):
- Belgium (2):
  - Novellas Healthcare, Asse
  - Associatie Orthopedie Hasselt, Hasselt

IPD SHARING:
Plan to Share IPD: No